CLINICAL TRIAL: NCT00590148
Title: Assessing Function in Pediatric Patients With Sickle Cell Disease Hospitalized With Vasoocclusive Pain Using the FIM Instrument
Brief Title: Assessing Function in Pediatric Patients With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, William Zempsky, MD, Director, Pain Relief Program, Connecticut Children's Medical Center
Other Study IDs: 07-163
Record Dates: First submitted 2007-12-27; First posted 2008-01-10 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the FIM™ as a measure of daily function in children with sickle cell disease hospitalized with vasoocclusive pain. Currently, the standard for pain assessment is a rating of pain intensity, as determined by observation (for younger children) or self-report (for older children and adolescents). However, these measures of pain intensity are not effective in recurrent or chronic pain states, and in sickle cell disease in particular. Pediatric patients who are hospitalized with vasoocclusive pain often do not report a decrease in pain intensity; however, other indications of clinical status, such as ambulation, less use of opiates from the patient-controlled analgesia (PCA) pump, increased food intake, and transition to oral pain medication, signify that the patient may be improving. As a result of our inability to get an accurate picture of the patients' condition, we would like to have a summary of improvement that would reflect these changes in clinical status and reflect the reduced impact of sickle cell pain on the patient's life. In this study, we plan to evaluate a standardized functional assessment measure in pediatric patients with sickle cell disease. It is hypothesized that FIM™ scores will correlate with other indicators of clinical status, such as movement, quality of sleep, use of IV opiates from the patient-controlled analgesia (PCA) pump, and use of intravenous vs. oral pain medications. It is also hypothesized that the FIM™ will demonstrate adequate responsiveness to change in functional status within a 3-7 day hospitalization by a progressive increase in scores and associations with other indicators of clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

* Ages 7-21 years inclusive
* Documented sickle cell disease
* Sudden onset of pain consistent with vasoocclusive episode
* Pain requiring hospitalization and placement on standard clinical guideline for management of acute pain in sickle cell disease
* Cognitive ability to report pain on a 0-10 Numerical Rating Scale (NRS)
* Parental consent and child assent

Exclusion Criteria:

* Younger than 7 years old
* Primary diagnosis other than vasoocclusive pain
* Concurrent Acute Chest Syndrome (ACS)

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with sickle cell disease
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
FIM score | Daily

SECONDARY OUTCOMES:
Adolescent Pediatric Pain Tool (APPT) body outline score | Daily

CONTACTS AND LOCATIONS:
Overall Officials: William T Zempsky, MD, Principal Investigator — Connecticut Children's Medical Center
Locations (2):
- United States (2):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Johns Hopkins University School of Medicine, Baltimore, Maryland